CLINICAL TRIAL: NCT04609046
Title: Phase I Trial of Methotrexate, Rituximab, Lenalidomide, and Nivolumab (Nivo-MR2) Induction Followed by Lenalidomide and Nivolumab Maintenance in Primary CNS Lymphoma
Brief Title: Testing the Addition of Lenalidomide and Nivolumab to the Usual Treatment for Primary CNS Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-08331; NCI-2020-08331 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A051901 (Other: Alliance for Clinical Trials in Oncology); A051901 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2020-10-29; First posted 2020-10-30 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Primary Diffuse Large B-Cell Lymphoma of the Central Nervous System
MeSH Terms: interventions — Biopsy; Lenalidomide; Spinal Puncture; Magnetic Resonance Spectroscopy; Methotrexate; merphos; Nivolumab; Rituximab; CT-P10; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (rituximab, methotrexate, lenalidomide, nivolumab) (Experimental): INDUCTION: Patients receive rituximab IV on day 1, methotrexate IV over 2 hours or PO on day 2, lenalidomide PO daily on days 5-9, and nivolumab IV over 30 minutes on day 14. (In dose level IV that includes nivolumab, the doses of rituximab for cycles 2-6 may be given on the same day as nivolumab for the previous cycle). Treatment repeats every 14 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response, partial response, or stable disease proceed to maintenance therapy.
  MAINTENANCE: Within 6 weeks after the last dose of lenalidomide in induction therapy, patients receive lenalidomide PO daily on days 1-21, and nivolumab IV over 30 minutes on day 1. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Patients also undergo MRI, CT, PET/CT, lumbar puncture, bone marrow aspirate and biopsy, testicular ultrasound and ECHO. (See Detailed Description)
  Interventions: Procedure: Bone Marrow Aspiration and Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Lenalidomide; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Drug: Methotrexate; Biological: Nivolumab; Procedure: Positron Emission Tomography; Biological: Rituximab; Procedure: Ultrasound Imaging

INTERVENTIONS:
Procedure: Bone Marrow Aspiration and Biopsy — Undergo bone marrow aspirate and biopsy
Procedure: Computed Tomography — Undergo CT and PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Methotrexate — Given IV or PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
Procedure: Ultrasound Imaging — Undergo testicular ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This phase I trial tests the safety, side effects, best dose and effectiveness of lenalidomide when added to nivolumab and the usual drugs (rituximab and methotrexate) in patients with primary central nervous system (CNS) lymphoma. Lenalidomide may stop or slow primary CNS lymphoma by blocking the growth of new blood vessels necessary for tumor growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of cancer cells to grow and spread. Rituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Methotrexate is frequently combined with other chemotherapy agents to improve response. This study may help increase the understanding of lenalidomide and nivolumab use in primary CNS lymphoma treatment. In addition, it may help researchers see whether the control of CNS lymphoma can be extended by using these study drugs as maintenance (prolonged therapy) after control is achieved with the initial chemotherapy regimen (induction).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of lenalidomide when given in combination with high dose-methotrexate (HD-MTX) and rituximab, with or without nivolumab, as induction treatment of primary CNS lymphoma.

II. Determine the proportion of patients who are able to stay on maintenance therapy with lenalidomide and/or nivolumab for 6 months after induction treatment of primary CNS lymphoma.

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate (ORR) of the combination of methotrexate, rituximab, lenalidomide, nivolumab.

II. To evaluate the effect of the treatment regimen and lenalidomide / nivolumab maintenance on progression free survival (PFS).

III. To evaluate the effect of the treatment regimen and lenalidomide / nivolumab maintenance on overall survival (OS).

EXPLORATORY OBJECTIVES:

I. To analyze tumor tissue and cerebrospinal fluid (CSF) for gene expression profiles, and to correlate these profiles with treatment outcomes.

II. To determine whether CSF proteome and metabolome are predictors of outcomes (prognostic marker).

III. To assess response to therapy and minimal residual disease via MRI-based metrics and minimal residual disease of blood and CSF.

IV. To evaluate the relationship between neurocognitive deficits and tumor and brain volumetrics, as assessed by magnetic resonance imaging (MRI) and tumor metabolism.

OUTLINE: This is a dose-escalation study of lenalidomide.

INDUCTION: Patients receive rituximab intravenously (IV) on day 1, methotrexate IV over 2 hours or orally (PO) on day 2, lenalidomide PO daily on days 5-9, and nivolumab IV over 30 minutes on day 14. (In dose level IV that includes nivolumab, the doses of rituximab for cycles 2-6 may be given on the same day as nivolumab for the previous cycle). Treatment repeats every 14 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve complete response, partial response, or stable disease proceed to maintenance therapy.

MAINTENANCE: Within 6 weeks after the last dose of lenalidomide in induction therapy, patients receive lenalidomide PO daily on days 1-21, and nivolumab IV over 30 minutes on day 1. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

Patients also undergo magnetic resonance imaging (MRI) throughout the trial, computed tomography (CT) and positron emission tomography (PET)/CT during screening, and lumbar puncture at the end of the 6th cycle of induction, and after 6 months of maintenance. Patients may also undergo bone marrow aspirate and biopsy, testicular ultrasound and/or echocardiogram (ECHO) during screening.

After completion of study treatment, patients are followed up every 3 months for 2 years, then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven primary CNS diffuse large b-cell lymphoma confirmed by one of the following:

  * Brain biopsy or resection
  * Cerebrospinal fluid
  * Vitreous fluid
* No prior organ transplantation to exclude post-transplant lymphoproliferative disorders
* No prior chemotherapy or radiation therapy for lymphoma
* No prior allogeneic stem cell transplantation
* Use of systemic corticosteroids (dexamethasone up to 24 mg/day or equivalent) for disease control or improvement of performance status to be tapered as fast as clinically safe after initiation of therapy is permissible
* Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown and an agent that has known genotoxic, mutagenic and teratogenic effects. Therefore, female of childbearing potential (FCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) =< 7 days prior to registration
* Age >= 18 years
* Karnofsky performance scale (KPS) >= 40 (>= 50 for patients older than 60 unless related to lymphoma on investigator's opinion)
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Calculated creatinine clearance >= 50 mL/min by Cockcroft-Gault formula
* Total Bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* No evidence of non-Hodgkin's lymphoma (NHL) outside CNS
* No prior history of NHL
* No history of autoimmune disorder. Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as Systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (except short course of systemic corticosteroids for disease control or improvement of performance status or other immunosuppressive medications within 14 days prior to registration. Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if < 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study
* No prior or concurrent malignancies with exception of surgically cured carcinoma in situ (CIS) of the uterus, carcinoma of the skin without evidence of disease for >= 5 years
* No concurrent malignancy requiring active therapy
* No untreated hepatitis C virus (HCV) infection with detectable HCV viral load
* No untreated chronic hepatitis B virus (HBV) infection with detectable HBV viral load
* No untreated human immunodeficiency virus (HIV) infection or with detectable viral load or with CD4+T-cell count of less than 500/mm^3
* No history of HIV infection and evidence of Epstein Barr virus (EBV)-related primary central nervous system lymphoma (PCNSL)
* Inability to tolerate anticoagulation with acetylsalicylic acid, warfarin, or direct oral anticoagulants
* No other investigational agent
* No history of severe hypersensitivity reaction to any monoclonal antibody
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to or other agents used in study
* Sulfonamide drugs, trimethoprim, salicylates, nonsteroidal anti-inflammatory drugs, penicillin, vitamin C, ciprofloxacin, and proton pump inhibitors should be held at least 48 hours prior to methotrexate administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2021-05-24 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | During the first 14-day cycle of treatment
  Defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients (at least 2 of a maximum of 6 new patients). The number and severity of all adverse events will be tabulated and summarized in this patient population both overall and by dose level according to the Common Terminology Criteria for Adverse Events (CTCAE) Cancer Therapy Evaluation Program version 5.0 criteria. The grade 3+ adverse events will also be described and summarized in a similar fashion. This will provide an indication of the level of tolerance for this treatment combination in this patient group.
Proportion of evaluable patients who are able to stay on maintenance therapy | Up to 6 months
  The proportion of evaluable patients who meet the criteria for maintenance feasibility, along with the 95% exact binomial confidence interval, will be provided.

SECONDARY OUTCOMES:
Overall response | Up to 5 years
  Will be estimated by the number of patients with the objective status of complete response, unconfirmed complete response, or partial response divided by the total number of evaluable patients. The overall response rate with an exact binomial 95% confidence interval will be provided and will be analyzed at the end of induction therapy and again after all therapy (induction and maintenance).
Progression free survival (PFS) | Time from start of induction treatment to progression or death due to any cause
  The distribution of progression-free survival will be estimated using the method of Kaplan-Meier (Kaplan-Meier, 1958). PFS time from start of maintenance therapy will also be reported in a similar fashion as the PFS time starting from induction therapy.
Overall Survival (OS) | Time from start of induction treatment to death due to any cause
  The distribution of overall survival will be estimated using the method of Kaplan-Meier (Kaplan-Meier, 1958). OS time from start of maintenance therapy will also be reported in a similar fashion as the OS time starting from induction therapy.
Incidence of adverse events | Up to 5 years
  Toxicity will be measured by the CTCAE version 5.0. The maximum grade, frequency, and severity for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration and analyzed descriptively.

OTHER OUTCOMES:
Minimal residual disease (MRD) | Up to 5 years
  Will estimate the proportion of patients with MRD at each time point with 95% confidence intervals. Will also use swimmer plots and other graphical analyses to visualize when MRD is detected/not detected in sequential samples relative to progression of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro J Alencar, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (54):
- United States (54):
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - University of Miami Sylvester Comprehensive Cancer Center at Sole Mia, North Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - UI Healthcare Mission Cancer and Blood - Fort Dodge, Fort Dodge, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Hickman Cancer Center, Adrian, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Overlook Hospital, Summit, New Jersey
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm